CLINICAL TRIAL: NCT01013857
Title: Treating to Target for Patients With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H40013-33128-02
Record Dates: First submitted 2009-11-12; First posted 2009-11-16 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health coaching (Active Comparator): Phone patients every week to discuss medication adherence
  Interventions: Behavioral: Health coaching
- Health coaching plus home-titration (Experimental): Health coaches call patients every week to discuss medication adherence and to intensify medications if appropriate according to physician-created algorithm
  Interventions: Behavioral: Health coaching plus home titration

INTERVENTIONS:
Behavioral: Health coaching — Calling patients every week to discuss medication adherence
  Arms: Health coaching
Behavioral: Health coaching plus home titration — Calling patients every week and intensifying medications if appropriate based on physician-created algorithm
  Arms: Health coaching plus home-titration

SUMMARY:
Patients with poorly controlled hypertension will have improved hypertensive control with telephone coaching and with telephone coaching combined with home-titration of medications.

DETAILED DESCRIPTION:
Patients with poorly controlled hypertension are randomized to a control arm which receives telephone coaching or an active arm which receives telephone coaching plus intensification of medications via telephone coaching with the coaches using treatment algorithms approved by the patients' physician. These patients' blood pressure control will be compared with usual care patients in a passive arm (chart review only).

ELIGIBILITY:
Inclusion Criteria:

* 2 blood pressure readings above 145/90.

Exclusion Criteria:

* Cognitive impairment,
* Short life expectancy,
* Creatinine greater than 1.5,
* Inability to check blood pressures at home.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2009-01; Primary Completion 2010-02 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | 6 months

SECONDARY OUTCOMES:
Diastolic blood pressure | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bodenheimer, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Derived] Bennett H, Laird K, Margolius D, Ngo V, Thom DH, Bodenheimer T. The effectiveness of health coaching, home blood pressure monitoring, and home-titration in controlling hypertension among low-income patients: protocol for a randomized controlled trial. BMC Public Health. 2009 Dec 10;9:456. doi: 10.1186/1471-2458-9-456. PMID 20003300